CLINICAL TRIAL: NCT03294200
Title: Clinical Trial Evaluation of the Percutaneous 4Tech TriCinch Coil Tricuspid Valve Repair System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As per sponsor
Sponsor: 4Tech Cardio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 2101-01
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tricinch Coil System treatment (Experimental)
  Interventions: Device: TriCinch Coil System implantation

INTERVENTIONS:
Device: TriCinch Coil System implantation — Patients enrolled in this study with all eligibility criteria confirmed will be implanted with the TriCinch Coil System. This device offers a percutaneous treatment (access through the vein at the groin) to treat the leaking tricuspid valve, without the need for surgical intervention.

SUMMARY:
The objective of the study is to generate safety and performance data for the 4Tech TriCinch Coil System in symptomatic patients suffering from significant functional tricuspid regurgitation with annular dilatation.

The TriCinch Coil System is a percutaneous catheter-based medical device for tricuspid valve repair.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe functional tricuspid regurgitation (TR) defined as: TR severity 2+ to 4+ (according to semi-quantitative echocardiographic color flow doppler evaluation); and Annular diameter ≥ 40 mm confirmed by echocardiography
2. ≥ 18 years old
3. Subject has read and signed the informed consent prior to study related procedures.
4. Willing and able to comply with all required follow-up evaluations and assessments.
5. The 'Heart Team' assessment recommends TriCinch Coil Implantation
6. New York Heart Associate Classification ≥ II.
7. Left Ventricular Ejection Fraction ≥ 30%.
8. Heart failure symptoms (such as fluid retention and severe oedema, liver stasis) despite on optimized medical therapy by the local heart team; at minimum subject on diuretic use
9. Subject has suitable anatomy for investigational device implantation as per imaging requirements

Exclusion Criteria:

1. Currently participating in another investigational drug or device study.
2. Subject with Systolic pulmonary arterial pressure (sPAP) > 60mmHg as measured by Transthoracic Echocardiography (TTE)
3. Subject requiring another cardiac procedure in the framework of the index procedure; subject requiring a percutaneous procedure within 30 days before or after the procedure or a cardiac surgical procedure within 3 months before or after the procedure
4. Moderate or Severe tricuspid valve stenosis (defined as a mean gradient ≥5 mmHg at normal heart rate)
5. Aortic, mitral and/or pulmonic valve stenosis and/or regurgitation more than or equal to moderate
6. Mitral valve stenosis and/or regurgitation more than moderate
7. Intra-cardiac thrombus, mass or vegetation requiring active treatment.
8. Implanted inferior vena cava (IVC) filter.
9. Prior tricuspid repair or tricuspid replacement
10. Known allergy to contrast media, silicone, PET, Co-Cr, stainless steel or nitinol that cannot be adequately pre-medicated
11. History of cardiac transplantation
12. Contraindication to Transthoracic/Transoesophageal Echocardiography (TTE/TOE).
13. Endocarditis or severe infection within 12 months of scheduled implant procedure
14. Myocardial Infarction (MI) or known unstable angina within the 30 days prior to the index procedure
15. Cerebro Vascular Accident within the previous 6 months
16. Hemodynamic instability or on IV inotropes
17. Contraindication to anticoagulant therapy and antiplatelet therapy
18. Bleeding disorders or hypercoagulable condition (at risk of blood clots)
19. Active peptic ulcer or active GI bleeding within 3 months of scheduled implant procedure
20. Severe renal impairment or on dialysis
21. Life expectancy less than 12 months.
22. Acute anemia
23. Chronic Oral Steroid Use ≥ 6 months
24. Pregnant or lactating female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure
25. Pulmonary embolism within the last 6 months
26. Tricuspid Valve Tethering distance > 10 mm
27. Presence of trans-tricuspid pacemaker or defibrillator leads which are determined as immobile or interfering with the procedure, as evaluated by echocardiography.
28. Contra-indicated for blood transfusion or refuses transfusion
29. Patient undergoing emergency treatment
30. Patient without appropriate venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
All-cause mortality of the Per Protocol cohort at 30 days post procedure. | 30 days post procedure

SECONDARY OUTCOMES:
Number of individual adverse events related to the system or procedure. | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure
Echocardiographic changes compared to Baseline by means of echocardiographic semi-quantitative and quantitative measures | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure
Functional changes as compared to Baseline for New York Heart Association (NYHA) classification | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure
Rate of Heart Failure event post-procedure defined as a heart failure hospitalization or a heart failure hospitalization equivalent | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure
Exercise tolerance (Six Minute Walk Test) | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure
Quality of Life evaluation (Kansas City Cardiomyopathy Questionnaire). | 30 days, three (3), six (6), twelve (12) and twenty-four (24) months post procedure

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (3):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Monash Heart, Clayton, Victoria
- AZ Sint Jan Brugge-Oostende AV, Bruges, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Clinique Pasteur, Toulouse, France
- CardioVascular Center Frankfurt, Frankfurt am Main, Germany
- Netherlands (2):
  - St Antonius Hospital, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- United Kingdom (4):
  - Brighton & Sussex University Hospitals - Sussex County Hospital, Brighton
  - Leeds General Infirmary, Leeds
  - Kings College Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided